CLINICAL TRIAL: NCT06192030
Title: Machine Learning-based Model for Prediction of Survival and Mutations in Ovarian Metastases of Colorectal Cancer
Brief Title: Machine Learning Predicts Survival and Mutations in Ovarian Metastases of Colorectal Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Other Study IDs: wanghm7
Record Dates: First submitted 2023-10-09; First posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Ovarian Metastases of Colorectal Cancer
Keywords: Krukenberg tumor
MeSH Terms: conditions — Krukenberg Tumor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Primary tumor, metastatic tissue and normal tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective cohort: The cohort was retrospectively enrolled in The Sixth Affiliated Hospital, Sun Yat-sen University from August 2010 to August 2022. It is a training cohort.
  Interventions: Other: Prediction model
- Prospective cohort: The same inclusion/exclusion criteria were applied for the same center prospectively. It is a validation cohort.
  Interventions: Other: Prediction model

INTERVENTIONS:
Other: Prediction model — We develop and validate clinical models to predict patient survival and gene signatures in ovarian metastases of colorectal cancer.

SUMMARY:
The study aimed to develop and validate models to predict survival outcome and key mutations in patients with ovarian metastases of colorectal cancer, as well as to compare the differential gene expression between long-survival group and short-survival group.

DETAILED DESCRIPTION:
The investigator performed a retrospective-prospective cohort study with the aim of developing and validating comprehensive models to predict survival outcome and key mutations from multimodality data in patients with ovarian metastases of colorectal cancer. Secondly, the investigator aimed to compare the differential gene expression between long-survival group and short-survival group.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed colorectal cancer
* Unilateral or bilateral ovarian masses confirmed by peroperative imaging examination
* Patient requiring resection of their ovarian and/or peritoneal carcinomatosis
* 18 ≤ Age ≤ 85
* World Health Organization performance status ≤ 1
* Life expectancy > 12 weeks
* Adequate haematological, liver and renal function
* Patient information and signature of the informed consent form before the start of any treatment procedures

Exclusion Criteria:

* Ovarian metastases of origin other than colorectal
* Primary ovarian tumor
* Clinical data missing

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ovarian metastases from colorectal cancer
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-08-27 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Overall survival | At least 3-year follow up
  Overall survival was defined as the time from surgery to death, or to the last follow-up.
Disease-free survival | At least 1-year follow up
  Disease-free survival was defined as the interval between surgery and the first peritoneal or distant relapse or death from any cause.
Peritoneal-free survival | At least 1-year follow up
  Peritoneal-free survival was defined as the interval between surgery and the first peritoneal relapse. Ovarian metastasis has been shown to be a subtype of peritoneal metastasis.

SECONDARY OUTCOMES:
Rates of key gene mutation | At least 1-year follow up
  Rates of key gene mutation, such as microsatellite instability-high/DNA mismatch repair

CONTACTS AND LOCATIONS:
Locations (1):
- Sixth Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided